CLINICAL TRIAL: NCT00693082
Title: Polycystic Ovarian Syndrome: Impact of Flaxseed Supplementation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: recruitment and pilot funding issues
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00000854
Record Dates: First submitted 2008-06-03; First posted 2008-06-06 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2012-11

CONDITIONS: Polycystic Ovarian Syndrome
Keywords: PCOS; flaxseed
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Linseed Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Dietary Supplement: flaxseed

INTERVENTIONS:
Dietary Supplement: flaxseed — 1 tablespoon a day for first three days, increasing to two tablespoons a day for the next three days. On the 7th day start with 3 tablespoons per day and maintain dose throughout the duration of the study (11 weeks).

SUMMARY:
The overall aim of this study is to explore the effects of flaxseed supplementation and determine whether it is a feasible and potentially effective dietary intervention among women with polycystic ovarian syndrome (PCOS). Women, ages 18-45, with clinically confirmed PCOS (N=20) will be scheduled for baseline measures and then instructed and given supplies necessary to follow a flaxseed supplemented (30 g/day) diet for a period of three months, whereupon follow-up measures will be taken. Subjects will be asked to resume their typical (unsupplemented) diet for another three months and a second set of follow-up measures will be taken. Baseline levels of bioavailable and total testosterone, fasting insulin, glucose, and triglycerides (TG), total/LDL/HDL cholesterol, body weight, degree of hirsutism and acne, and menstrual cyclicity will be compared to levels at 3 and 6 month follow-up. The overall hypothesis (based upon our work in men at risk for prostate cancer and data from one case-study conducted in a woman with confirmed PCOS) is that during the time women receive flaxseed supplementation they will experience reduced serum levels of testosterone, and total and LDL cholesterol, as well as clinical evidence of hirsutism. Given the pilot nature of this study, statistical analyses will be limited to simple descriptive statistics. We have observed no negative side effects, other than minor gastro-intestinal occurrences (i.e., temporary increased flatulence, borborygmi, increased number of stools, etc.) associated with flaxseed supplementation in our previous studies either with short or long-term use. Flaxseed supplementation will be discontinued if indicated and the events reported to the institutional review board.

ELIGIBILITY:
Inclusion Criteria:

* limited to women aged 18-45
* diagnosis of PCOS by menstrual irregularity (fewer than 9 menses annually), Ferriman-Gallwey score > 8, and/or hyperandrogenemia defined as bioavailable T>8.4ng/dL (Zawdaki & Dunaif 1992)
* mentally competent
* English speaking/writing
* telephone access and/or email access

Exclusion Criteria:

* Use of oral contraceptives, spironolactone or insulin-sensitizing agents within the past 3 months;
* Long-term or chronic use of oral antibiotics;
* Diagnoses of hyperprolactinemia, thyroid abnormalities, or nonclassic adrenal hyperplasia;
* Hysterectomy;
* Onset of menopause;
* Pregnancy/Lactation;
* Consumption of flaxseed within the past month; and
* Use of any dietary fiber supplements which are newly started (within the past 6 months) and agreement not to use any new fiber supplements during the study period

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2007-08; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
To explore the effects of flaxseed supplementation on women with clinically confirmed PCOS. | baseline, 12 weeks, 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Susan M Schneider, PhD, Principal Investigator — Duke University
Locations (1):
- Duke Univeristy Medical Center, Durham, North Carolina, United States